CLINICAL TRIAL: NCT05697276
Title: Which Combination of Local Anesthesia is Superior for Postoperative Pain After Carpal Tunnel Surgery?: A Prospective Randomized Study.
Brief Title: Are There Differences in Postoperative Pain Between Bupivacaine and Lidocaine for Carpal Tunnel Release?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Italiano de Buenos Aires (Other)
Responsible Party: Principal Investigator, IGNACIO RELLAN, Principal investigator, Hospital Italiano de Buenos Aires
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 6337
Record Dates: First submitted 2022-12-31; First posted 2023-01-25 (Actual); Last update posted 2023-08-29 (Actual); Status verified 2023-08

CONDITIONS: Carpal Tunnel Syndrome; Carpal Tunnel
Keywords: Carpal Tunnel Syndrome; Postoperative Pain; Bupivacaine; WALANT; Lidocaine
MeSH Terms: conditions — Carpal Tunnel Syndrome; Median Neuropathy; Pain, Postoperative | interventions — Lidocaine; Bupivacaine

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lidocaine (Active Comparator): Patients will receive lidocaine
  Interventions: Drug: Lidocaine
- Bupivacaine (Experimental): Patients will receive bupivacaine
  Interventions: Drug: Bupivacain

INTERVENTIONS:
Drug: Lidocaine — Patients will receive 20 ml of 1% lidocaine with 1:100,000 epinephrine (buffered 10:1 with 8.4% sodium bicarbonate). Thirty minutes before carpal tunnel release surgery, 10 mL will be injected subcutaneously, and 10 mL will be injected into the carpal tunnel.
  Arms: Lidocaine
Drug: Bupivacain — Bupivacaine: Patients will receive 10 ml of 0.5% bupivacaine + 10 ml of 1% lidocaine with 1:100,000 epinephrine (buffered 10:1 with 8.4% sodium bicarbonate). Thirty minutes before carpal tunnel release surgery, 10 mL will be injected subcutaneously, and 10 mL will be injected into the carpal tunnel.
  Arms: Bupivacaine

SUMMARY:
The goal of this clinical trial is to compare the use of bupivacaine and lidocaine as local anesthetics in carpal tunnel release surgery. The main questions it aims to answer are:

* Are there any differences in pain after surgery?
* Are there any differences in postoperative analgesic consumption?

DETAILED DESCRIPTION:
The Wide-Awake Local Anesthesia No Tourniquet (WALANT) technique has become popular for hand surgery in the past decade. It consists of injecting a local anesthetic and epinephrine into the surgical site. Lidocaine, a short-acting local anesthetic, is used in the classic description. Adding a long-acting local anesthetic, such as bupivacaine, has been suggested for long surgeries.

However, the use of bupivacaine in shorter-duration procedures could combine the advantages of ambulatory surgery without a tourniquet with long-acting analgesia, improving postoperative pain and reducing the consumption of analgesics.

Patients undergoing first-time open carpal tunnel release surgery will be randomized to receive bupivacaine or lidocaine. Randomization will be generated by computer using random block sizes of 2 or 4 with an allocation ratio of 1:1.

Postoperatively, patients will receive standard medical care. It consists of 50 mg of diclofenac to take when they feel pain (with a minimum interval of 8 hours). Patients will be instructed to complete a medication log for pain and analgesic consumption. A blinded investigator will contact them by phone at 24 hours and 48hs. At two weeks, they will be controlled by research staff for complications.

Eighty-two patients will be recruited, 41 per arm, assuming a 20% loss. The sample size was calculated using a 90% power and 5% significance level. The objective was to detect a minimum difference of 2 points on a numeric scale ranging from 0 to 10 with a standard deviation of 2.5 points.

ELIGIBILITY:
Inclusion Criteria:

* Patients with carpal tunnel syndrome undergoing first-time surgery

Exclusion Criteria:

* Pregnant
* End-stage kidney disease
* End-stage liver disease
* Allergy to bupivacaine, lidocaine or diclofenac
* Carpal tunnel revision surgery
* Associated surgery (e.g., trigger finger release)
* Unable to understand informed consent or indications
* Patients with anxiety related to surgery who explicitly prefer to be sedated or asleep during their surgery
* Preoperative American Society of Anaesthesiology (ASA) scale ≥3

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2022-09-13 (Actual); Primary Completion 2023-08-07 (Actual); Study Completion 2023-08-26 (Actual)

PRIMARY OUTCOMES:
Postoperative Pain | Change in pain at 24 and 48 hours or when the patients take analgesics
  Visual analog scale, numerical scale from 0 to 10
Time until pain | Until 48 hours from surgery
  Time in hours (numeric) from surgery until the patient feel pain
Amount of analgesic | at 24 and 48 hours
  The number of analgesics consumed by the patient. Numeric

SECONDARY OUTCOMES:
Pain during anesthesia | 1 minute after the injection of local anesthesia
  Visual analog scale, numerical scale from 0 to 10
interruption of sleep due to pain | at 24 hours
  Did the patient wake up because of pain the first night?, Categorical, Yes or No

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital italiano de Buenos Aires, Buenos Aires, Other, Argentina

REFERENCES:
- [Background] Lalonde D, Martin A. Epinephrine in local anesthesia in finger and hand surgery: the case for wide-awake anesthesia. J Am Acad Orthop Surg. 2013 Aug;21(8):443-7. doi: 10.5435/JAAOS-21-08-443. PMID 23908250
- [Background] Lalonde DH. "Hole-in-one" local anesthesia for wide-awake carpal tunnel surgery. Plast Reconstr Surg. 2010 Nov;126(5):1642-1644. doi: 10.1097/PRS.0b013e3181f1c0ef. No abstract available. PMID 21042120
- [Background] Lalonde D. Minimally invasive anesthesia in wide awake hand surgery. Hand Clin. 2014 Feb;30(1):1-6. doi: 10.1016/j.hcl.2013.08.015. Epub 2013 Nov 9. PMID 24286736
- [Background] Chan ZH, Balakrishnan V, McDonald A. Short versus long-acting local anaesthetic in open carpal tunnel release: which provides better preemptive analgesia in the first 24 hours? Hand Surg. 2013;18(1):45-7. doi: 10.1142/S0218810413500081. PMID 23413849
- [Background] Diaz-Abele J, Luc M, Dyachenko A, Aldekhayel S, Ciampi A, McCusker J. Lidocaine With Epinephrine Versus Bupivacaine With Epinephrine as Local Anesthetic Agents in Wide-Awake Hand Surgery: A Pilot Outcome Study of Patient's Pain Perception. J Hand Surg Glob Online. 2019 Oct 31;2(1):1-6. doi: 10.1016/j.jhsg.2019.09.004. eCollection 2020 Jan. PMID 35415474